CLINICAL TRIAL: NCT06433024
Title: A Pilot Study Using AI Algorithms and PPG Technology for the Detection of Venous Diseases
Brief Title: Training of a Artificial Intelligence Model to Detect Venous Diseases Using PPG Technology
Status: Not yet recruiting | Type: Observational
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: TWC-SD-2024-05
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Venous Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Individuals with CVD (Treatment Group): Participants who have been diagnosed with Chronic Venous Disease (CVD).
  Interventions: Diagnostic Test: PPG Diagnostic
- Individuals Without CVD (Control Group): Participants who have not been diagnosed with CVD.
  Interventions: Diagnostic Test: PPG Diagnostic

INTERVENTIONS:
Diagnostic Test: PPG Diagnostic — The study investigates venous competence through three distinct exercises using photoplethysmography (PPG) technology to record blood flow in the leg veins of 20 subjects, split into two groups: those with chronic venous disease (CVD) and those without. The null hypothesis is that there will be no significant difference in venous filling times (VFT) and PPG trace variations between subjects with CVD and those without under different physical conditions. The alternative hypothesis suggests that individuals with CVD will show distinct PPG patterns, particularly shorter VFT and varied pressure changes, indicative of venous reflux or obstruction. This hypothesis is chosen based on prior evidence suggesting observable differences in venous function between affected and non-affected individuals.

SUMMARY:
This clinical research aims to evaluate the effectiveness of using Photoplethysmography (PPG) signals combined with Artificial Intelligence (AI) algorithms, for the precise classification and diagnosis of Venous Diseases of the lower limb. This study invites a group of participants who currently undergoing investigations for venous disease at The Whiteley Clinic (hereinafter referred to as TWC). The Participants will be classified into control (healthy individuals with no significant venous disease) and chronic venous disease (CVD) (diagnosed with proven venous disease) groups. Prospective participants who express an interest in being included in the study will be given a patient information sheet and will undergo a briefing of the pilot study. If they consent and sign the relevant consent forms, the participants will perform a series of standardized exercises under the supervision of a consultant vascular surgeon. Throughout the exercises, a data acquisition device attached to the ankle records the PPG signals, capturing the changes in blood volume due to the reflected PPG signals from the red blood cells during the movement. Thus, once the data is collected and recorded, this allows for the analysis of the data of the control group and CVD group against each other. During the analysis of the two groups' PPG signals, the objective lies within the capability to detect subtle nuances in the patterns of the PPG signals during the performed movements using AI algorithms. The AI algorithms will distinguish patterns or features indicating the presence or absence of venous disease. This study seeks to contribute valuable insights into enhancing the diagnosis of venous disease using PPG and AI algorithms, paving novel approaches to Venous healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Patients are attending for investigation of suspected venous disease. Patients must be able to walk and mobile normally and have good skin integrity of the lower leg, where the PPG is attached.

All patients attending TWC are 18 years or older.

Exclusion Criteria:

* Subjects with known arterial occlusive disease or physical disability affecting gait or ankle movement will be excluded.

Patients unable to have a PPG attached to the lower leg (ie: active ulceration) will be excluded.

Patients unable to give consent. Pregnant female.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study invites a group of participants who have attended The Whiteley Clinic (hereinafter referred to as TWC). The Participants are split into control (healthy individuals) and treatment (previously diagnosed with Venous disease) groups.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of an AI Model for Venous Disease Detection Using PPG Signals | June 2024 - September 2024
  The primary outcome measure of this study is to evaluate the diagnostic accuracy of an AI model in detecting venous disease through the using PPG signals. This will be quantified by assessing the sensitivity and specificity of the AI model when analysing PPG signals from healthy participants without venous diease, and non-healthy participants with venous disease, without the need for direct intervention of a vascular consultant. These results will help evaluate the AI model in terms of how accurately it can identify Venous disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Whiteley, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No